CLINICAL TRIAL: NCT03452436
Title: Testosterone, Cognition, Ageing, and Cancer - A Controlled, Prospective Study About the Association Between Testosterone and the Prevalence and Severity of Cancer Related Cognitive Impairment in Testicular and Prostate Cancer Patients.
Brief Title: Testosterone, Cognition, Ageing, and Cancer
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TCAC
Record Dates: First submitted 2018-02-01; First posted 2018-03-02 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-04

CONDITIONS: Cancer-related Cognitive Impairment
Keywords: Cancer-related Cognitive Impairment; Cognitive Dysfunction; Cognition Disorders; Neurocognitive Disorder; Testosterone; Endocrinology; Testicular Cancer; Prostate Cancer
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders; Neurocognitive Disorders; Testicular Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Testicular cancer patients: Forty testicular cancer patients included after orchiectomy but prior to any further treatment.
- Prostate cancer patients: Forty prostate cancer patients included prior to medical castration and radiotherapy.
- Healthy controls: Forty age- and education-matched healthy controls (20 matched to testicular cancer patients, 20 matched to prostate cancer patients).

SUMMARY:
The primary aim of the study is - in a prospective controlled design - to examine whether treatment-induced decreases in testosterone acts as a mechanism of cancer-related cognitive impairment (CRCI) in testicular and prostate cancer patients.

Secondary aims are 1) to explore whether decreases in testosterone interacts with increasing age to cause more severe CRCI in older patients, 2) to explore underlying neurophysiological (brain morphology) mechanisms of CRCI, and 3) to evaluate selected genetic variants as possible moderators of CRCI.

DETAILED DESCRIPTION:
The study will include three groups with a total of 120 participants: A) Forty testicular cancer patients will be included and examined 1) shortly after orchiectomy and prior to any further treatment and 2) at 6 months' follow- up. B) Forty prostate cancer patients will be included and examined at two time-points: 1) prior to initiation of medical castration and radiotherapy and 2) at 6 months' follow- up. C) Forty age- and education-matched healthy controls will be included and assessed at a similar time-interval, i.e., at an initial examination and at a 6 month follow-up. Measures include a battery of neuropsychological/ cognitive tests, questionnaires, blood samples, and Magnetic Resonance Imaging (MRI).

Primary hypothesis

1. Treatment-induced decreases in testosterone will be associated with decline in global cognitive functioning from baseline to 6 months' follow- up in both testicular and prostate cancer patients.

   Secondary hypotheses
2. Treatment-induced decreases in testosterone will be associated with decline in individual cognitive domains (i.e., processing speed, attention, verbal fluency, executive functioning, working memory, verbal learning and memory, visuospatial learning and memory, and visuospatial ability) from baseline to 6 months' follow- up in both testicular and prostate cancer patients.
3. Decline in cognitive functioning from baseline to 6 months' follow- up in both testicular and prostate cancer patients will correspond to changes in grey matter as measured by T1-weighted MRI.
4. Decline in cognitive functioning from baseline to 6 months' follow- up in both testicular and prostate cancer patients will correspond to changes in brain white matter as measured with diffusion-weighted MRI.
5. Treatment-induced decreases in testosterone will be more strongly associated with decline in cognitive functioning in prostate cancer patients compared with testicular cancer patients due to more advanced age in the former group.
6. Treatment-induced decreases in testosterone will be more strongly associated with decline in cognitive functioning in both testicular and prostate cancer patients carrying the the Apolipoprotein E (APOE) ε4 allele, the Val catechol-O-methyltranferase (COMT) allele, the Val/Val Brain- derived neurotrophic factor (BDNF) genotype, and a short polymorphic CAG repeat length of the Androgen Receptor (AR) gene.
7. Treatment-induced decreases in testosterone will be associated with increases in neurobehavioral symptoms (i.e., apathy, executive dysfunction, and disinhibition) from baseline to 6 months' follow- up in both testicular and prostate cancer patients.
8. Treatment-induced decreases in testosterone will be associated with decreases in health-related quality of life from baseline to 6 months' follow- up in both testicular and prostate cancer patients.
9. Treatment-induced decreases in testosterone will be associated with decreases in perceived cognitive functioning from baseline to 6 months' follow- up in both testicular and prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of testicular cancer
* Confirmed diagnosis of prostate cancer and prescription of medical castration and radiotherapy

Exclusion Criteria:

* Previous cancer disease
* Previous central nervous system disease
* Brain metastases
* Severe psychiatric disease (e.g., schizophrenia, major depressive disorder)
* Insufficient Danish proficiency for neuropsychological testing

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men with testicular and prostate cancer seen at Aarhus University Hospital. Age- and education matched healthy controls recruited from the general population of Central Denmark Region.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Global cognitive functioning | Baseline and 6 months' follow-up
  Changes in global cognitive composite score as measured with neuropsychological tests specified under "Secondary Outcome Measures".

SECONDARY OUTCOMES:
Visuospatial ability | Baseline and 6 months' follow-up
  Changes in visuospatial ability as measured with WAIS-IV Matrix Reasoning.
Visuospatial ability | Baseline and 6 months' follow-up
  Changes in visuospatial ability as measured with WAIS-IV Figure Weights.
Visuospatial ability | Baseline and 6 months' follow-up
  Changes in visuospatial ability as measured with WAIS-IV Visual Puzzles.
Visuospatial ability | Baseline and 6 months' follow-up
  Changes in visuospatial ability as measured with WAIS-IV Block Design.
Processing speed | Baseline and 6 months' follow-up
  Changes in processing speed as measured with Trail Making Test A.
Processing speed | Baseline and 6 months' follow-up
  Changes in processing speed as measured with WAIS-IV Coding.
Attention | Baseline and 6 months' follow-up
  Changes in attention as measured with WAIS-IV Digit Span Forwards.
Executive functioning | Baseline and 6 months' follow-up
  Changes in executive functioning as measured with Trail Making Test B.
Executive functioning | Baseline and 6 months' follow-up
  Changes in executive functioning as measured with Wisconsin Card Sorting Test.
Working memory | Baseline and 6 months' follow-up
  Changes in working memory as measured with WAIS-IV Digit Span Sequencing.
Working memory | Baseline and 6 months' follow-up
  Changes in working memory as measured with WAIS-IV Digit Span Backwards.
Verbal fluency | Baseline and 6 months' follow-up
  Changes in verbal fluency as measured with Controlled Oral Word Association Test.
Verbal learning and memory | Baseline and 6 months' follow-up
  Changes in verbal learning and memory as measured with Hopkins Verbal Learning Test-Revised.
Visuospatial learning and memory | Baseline and 6 months' follow-up
  Changes in visuospatial learning and memory as measured with WMS-III Visual Memory.
Testosterone levels | Baseline and 6 months' follow-up
  Changes in testosterone levels as measured with liquid chromatography tandem mass spectrometry (LC-MS/MS).
Brain grey matter | Baseline and 6 months' follow-up
  Changes in grey matter as measured with T1-weighted MRI.
Brain white matter | Baseline and 6 months' follow-up
  Changes in brain white matter as measured with diffusion-weighted MRI.
Moderator: APOE genotype | Baseline
  Genotype of the APOE gene obtained by TaqMan-genotyping the appropriate single nucleotide polymorphisms.
Moderator: COMT genotype | Baseline
  Genotype of the COMT gene obtained by TaqMan-genotyping the appropriate single nucleotide polymorphism.
Moderator: BDNF genotype | Baseline
  Genotype of the BDNF gene obtained by TaqMan-genotyping the appropriate single nucleotide polymorphism.
Moderator: CAG repeat length of the AR gene | Baseline
  CAG repeat lenght of the AR gene obtained by TaqMan-genotyping the appropriate single nucleotide polymorphism.
Neurobehavioral symptoms (i.e., apathy, executive dysfunction, and disinhibition) | Baseline and 6 months' follow-up
  Changes in neurobehavioral symptoms as measured with The Frontal Systems Behavior Scale (FrsBe).
Perceived cognitive functioning | Baseline and 6 months' follow-up
  Changes in perceived cognitive functioning as measured with The Patient Assessment of Own Functioning Inventory (POAFI).
Health-related quality of life | Baseline and 6 months' follow-up
  Changes in health-related quality of life as measured with The European Organization for Research and Treatment of Cancer, Quality of Life questionnaire for cancer patients (EORTC QLQ-C30).
Health-related quality of life - Prostate Cancer | Baseline and 6 months' follow-up
  Changes in disease specific health-related quality of life as measured with The European Organization for Research and Treatment of Cancer, Quality of Life Prostate Cancer Module (EORTC QLQ-PR25).
Health-related quality of life - Testicular Cancer | Baseline and 6 months' follow-up
  Changes in disease specific health-related quality of life as measured with The European Organization for Research and Treatment of Cancer, Quality of Life Testicular Cancer Module (EORTC QLQ-TC25).

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie D R Clausen, MSc, Principal Investigator — Unit for Psychooncology & Health Psychology, Department of Oncology, Aarhus University; Robert Zachariae, Professor, DMSc, Study Director — Unit for Psychooncology & Health Psychology, Department of Oncology, Aarhus University
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided